CLINICAL TRIAL: NCT04677634
Title: Open Label Tolerability Study of ISOThrive Prebiotic Nectar, Maltosyl-Isomalto-oligosaccharides (MIMO), in Subjects With Constipation
Brief Title: Open Label Tolerability Study of ISOThrive Prebiotic Nectar (MIMO) in Subjects With Constipation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ISOThrive Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1002
Record Dates: First submitted 2020-12-16; First posted 2020-12-21 (Actual); Last update posted 2022-05-05 (Actual); Status verified 2022-05

CONDITIONS: Constipation
Keywords: IBS-C; MIMO; remote
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tolerability Arm (Other): This is a single arm study. All subjects will receive the test material. The test material is ISOThrive. It is an approximately 90% pure maltosyl-isomalto-oligosacchride (MIMO) prebiotic syrup produced by bacterial fermentation/bio-conversion of sucrose and maltose. It is taken 1g daily for 30 days.
  Interventions: Dietary Supplement: ISOThrive Prebiotic Nectar

INTERVENTIONS:
Dietary Supplement: ISOThrive Prebiotic Nectar — The test material is ISOThrive. It is an approximately 90% pure maltosyl-isomalto-oligosacchride (MIMO) prebiotic syrup produced by bacterial fermentation/bio-conversion of sucrose and maltose. It is taken 1g daily.
  Other Names: ISOT-101; maltosyl-isomaltooligosaccharides; MIMO

SUMMARY:
The purpose and efficacy endpoint of this study is to assess whether subjects with constipation predominant irritable bowel syndrome (IBS-C) or chronic Idiopathic constipation (CIC) tolerate ISOThrive.

DETAILED DESCRIPTION:
Study Design The test material is ISOThrive. It is an approximately 90% pure maltosyl-isomalto-oligosacchride (MIMO) prebiotic syrup produced by bacterial fermentation/bio-conversion of sucrose and maltose. It is taken 1g daily.

Subjects will have been screened for CIC or IBS-C as determined by the Rome IV criteria during an interview with the study coordinator and by evaluation of the online questionnaire responses for PAC-QOL, PAC-SYM, and BSS. The study has been designed to have each subject serve as their own control so there will be no placebo arm. Each subject will receive ISOThrive according to the protocol. The goal is to assess 100 subjects after the Screening Phase. The study will be done remotely. There will be communication but no in person contact or visits with the study coordinator.

Two phases have been designed into this study. Phase 1 is the Screening Phase (SP) lasting 7 days. Phase 2 is the Tolerability Phase (TP) lasting 28 days. Subjects will be instructed to take a daily BSS questionnaire and bowel movement frequency throughout the study. They will note whether they have had bowel movements each day and describe them accordingly. At three timepoints, specific scores will be established for comparison and statistical analysis. These timepoints are: (1) SP7 - baseline without ISOThrive; (2) TP14 - 2 weeks using ISOThrive; (3) TP28 - 4 weeks using ISOThrive. At each of these timepoints, subjects will also complete the PAC-QOL and PAC-SYM validated questionnaires. Subjects will report any usage of laxatives and any changes in their usual medications throughout their study participation on a daily basis.

Enrollment An adequate number of individuals will need to be screened during the Screening Phase, using the disease specific validated questionnaires to yield approximately 100 qualified subjects to enter and likely complete the Tolerability Phase of the study. Individuals on medications for CIC or IBS-C may continue their medications during the trial as long as they are reported and do not deviate from the inclusion/exclusion criteria.

All subjects will be required to sign an IRB-approved informed e-consent that complies with the requirements of both 21 CRF Part 50 and Health Insurance Portability and Accountability Act (HIPAA) before entering the study.

The duration of the study is defined for each subject as the date a signed written informed consent (or e-consent) is provided through Tolerability Phase Day 28. Total participation in study may last up to 6 weeks. The study will seek a comparable gender distribution in the final analysis. Therefore, the ratio of male to female (or female to male) subjects completing the Tolerability Phase will be capped at 60% of the total (male or female).

Concomitant Medications and Washout Periods CIC and IBS-C medications: Subjects currently taking laxatives or other treatments for CIC or IBS-C may continue these throughout the study. These will be recorded. Any changes in dosing of these will also be recorded. Commercially available medications or supplements marketed as prebiotics or probiotic cannot be taken. Supplements such as Metamucil and Citrucel are acceptable in this study.

Prebiotic and/or probiotic supplements: Enrolled subjects must stop taking all prebiotic and/or probiotic supplements 3 weeks prior to entering the Screening Phase of the study. Subjects must refrain from taking prebiotic or probiotic supplements through Tolerability Phase Day 28.

Sleep medications: Enrolled subjects taking medications for mild sleep disorders must be on a stable dose at time of consent and continue at said dose through Tolerability Phase Day 28.

Antibiotics: Subjects must not have taken a 10 day course of a single antibiotic within the past 3 months, >10 day course of a single antibiotic during the past 5 months, course of >1 antibiotics within the past 5 months , or at any time during their participation in the study. If antibiotics are prescribed to the subject during study participation, subject must be withdrawn from study.

All study product sachets (used and unused) must be returned to Investigator for product accountability.

Subject Study Flow Process No study-related activities will be performed and no subject data will be collected prior to completion of the informed consent process.

Screening Phase (SP) (7 days):

To enter the SP, subjects must be screened for CIC or IBS-C during an interview with the study coordinator using the Rome IV criteria and also by the study questionnaires. The SP will last for 7 days. Subjects who do not qualify at any point during the SP will not be allowed to move into the Tolerability Phase (TP). The TP will last 28 days, beginning with first dose of ISOThrive. Subjects will continue their allowed CIC or IBS-C medications throughout the SP and the TP.

Following Day 7 of SP, a review of the questionnaire responses will be made. Subjects must complete at least 5 of 7 daily BSS questionnaires. Combined BSS, bowel movement frequency, PAC-QOL and PAC-SYM responses will be evaluated for consistency with CIC or IBS-C per the Rome IV criteria by the PI to be eligible to transition to the Tolerability Phase. (Two or fewer bowel movements in a week which resulted in a sensation of complete evacuation with one or more of the following: lumpy or hard stools at least 25% of the time, sensation of incomplete evacuation at least 25% of the time, sensation of anorectal obstruction or blockage for at least 25% of the time, manual maneuvering required to defecate for at least 25% of the time, or straining at defecation at least 25% of the time.) The PAC-QOL, PAC-SYM and BSS and bowel movement frequency scores will serve as a baseline. Investigator will verify eligibility prior to study staff contacting subject.

Once eligibility has been verified by the PI, the study coordinator will inform subject and confirm that subject wishes to continue in the study. There may be up to 7 calendar days between SP Day 7 and TP Day 1 depending on length of time to evaluate continuing eligibility and to ship/receive ISOThrive.

Tolerability Phase (TP) (28 days):

Subjects will take their current CIC or IBS-C therapy as defined in the inclusion/exclusion section.

All CIC or IBS-C medications and other medications will be recorded daily via the electronic survey.

ISOThrive will be taken daily each morning with or without breakfast (one sachet per day). If the subject forgets to take the morning dose, he/she may take it during the day or evening. If the dose is forgotten for 24 hours, the subject may take a double dose the next day. The product must be taken at least 6 of 7 days each week. Only 2 double doses per week are allowed (but discouraged).

As the primary endpoint, tolerability of ISOThrive will be assessed via changes in the BSS, bowel movement frequency, PAC-QOL, and PAC-SYM and questionnaires. This will be assessed for all subjects as well as for the sub-group of subjects that completed all 4 weeks of the TP. Changes in BSS (frequency and stool quality), PAC-QOL, or PAC-SYM, between baseline and each of the TP14 and TP28 time points will be the basis of this assessment. Subjects also rated the change in their constipation on a 7-point scale (very much improved to very much worsened) at the final follow-up (TP28). Further evaluation will include comparison of ISOThrive tolerability in CIC vs IBS-C subject sub-groups using these time points.

The safety endpoint of the study is to ensure that any adverse events that are reported or observed during the study are appropriately recorded.

Subject Reimbursement Except for a $25 gift card for completion of all study requirements, no additional study compensation is being given to the research participant or authorized representative for data collected from this study. All study participants will be provided with ISOThrive for the duration of their participation in the study.

Adverse Events Adverse events (AEs) may occur during the conduct of the study. As no changes to treatment plans will be made during the Screening Phase, AEs will be captured at the time of entry into the Tolerability Phase and continue through the last study conduct (TP Day 28) for each subject. AEs will be recorded in the case report forms and will be judged by the Investigator as to its relationship and level of relatedness to the study product. Investigator will identify the date of onset, severity, and duration of the AE. All AEs will be monitored until they are adequately resolved or explained. If an AE continues after the evaluation of the study, the Investigator will determine need and/or methods for continued surveillance of the event.

The Investigator will report adverse events and/or serious adverse events to the reviewing IRB according to the reporting regulations.

Data Quality Assurance This study will be conducted in accordance with the International Council for Harmonization (ICH) E6 R2. The Investigator agrees to maintain adequate documentation for the subjects participating in this clinical research project. The Investigator agrees to maintain accurate case report forms and source documentation as part of the case histories. Subjects will enter their data into the data capture system (REDCap). The analysis data sets will be generated from data captured in REDCap.

Ethical Considerations The rights, safety and wellbeing of clinical investigation subjects shall be protected consistent with the ethical principles outlined in the Declaration of Helsinki. This shall be understood, observed, and applied at every step in this clinical investigation.

Protection of Subject Confidentiality At all times throughout this clinical investigation, confidentiality will be observed by all parties involved. All data shall be secured against unauthorized access. Privacy and confidentiality of information about each subject shall be preserved in the reports and in any publication. Each subject participating in this study will be assigned a unique identifier. All CRFs will be tracked, evaluated, and stored using only this unique identifier.

Data Collection and Management Study data will be collected using standardized Case Report Forms (CRFs). The CRFs are designed to accommodate the specific features of the trial design. All data will be handled as applicable, per Good Clinical Practice. Data entry will be performed only by qualified personnel assigned by the Investigator. Passwords will be issued to appropriate personnel to ensure confidentiality and protection of data.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking male and female adults between the ages of 18 and 75, inclusive
2. Body mass index (BMI) <35 and >19, inclusive
3. IBS-C or CIC based on the Rome IV criteria (see Appendix 1) determined via phone interview with the study coordinator and via responses to the questionnaire responses during the Screening Phase
4. History (minimum of three months) of constipation as defined in appendix #1
5. Must be on stable doses of medications, if any, prescribed for chronic conditions other than IBS-C or CIC
6. If female of child-bearing age, must be on an active contraceptive measure or have male partner(s) with suitable protective measures
7. Have access to a computer/tablet/phone with internet access and active e-mail account to complete electronic surveys daily throughout study participation
8. Complete at least 5 of 7 daily BSS daily questionnaires and complete PAC-QOL and PAC-SYM questionnaires during the Screening Phase to enter the Tolerability Phase
9. Complete 5 of 7 BSS daily questionnaires each week and PAC-QOL and PAC-SYM questionnaires at the end of weeks 2 and 4 of the Tolerability Phase to remain in the study
10. Ability and willingness to give consent to participate in study

Exclusion Criteria:

1. Significant comorbidities that are not medically stable
2. History of any abdominal surgery involving the stomach, small or large intestine including appendectomy, cholecystectomy, pancreatic surgery, and any surgery involving abdominal trauma
3. History of diabetes (type I or type II)
4. History of any process that has resulted in abdominal adhesions, thus affecting gut motility
5. History of defecatory or rectal evacuation disorders, which may be based on specific tests such as colonic transition time, manometry evaluation and defecography, such as pelvic floor dyssynergia or a reduction in intra-abdominal pressure (act of bearing down), rectal sensory perception, and rectal contraction (Ohkusa et al. 2019)
6. History of diarrhea predominant or alternating diarrhea/constipation predominant IBS
7. BMI >=35, BMI <=19
8. Active history of nicotine use, cannabis use or alcohol abuse (as defined by: greater than 14 drinks/week or 4 drinks/day for men, 7 drinks/week or 3 drinks/day for women). Has used any tobacco, nicotine or cannabis products in the last 6 months or has abused alcohol in the last 6 months
9. Taking any opioids or any other constipating medications within the prior month
10. Must not take, and must not have taken within 3 weeks prior to commencing the Screening Phase, commercially available medications or supplements marketed as prebiotics or probiotics (Supplements such as Metamucil and Citrucel are acceptable in this study)
11. Having taken a 10 day course of a single antibiotic within the past 3 months, >10 day course of a single antibiotics during the past 5 months, or course of >1 specific antibiotic within the past 5 months;
12. Has any clinically significant finding which would confound the results, based on a physical exam or clinical laboratory testing after signing the consent but before receiving the first dose of study medication, based on determination by investigator;
13. Reports using a prohibited medication or dietary supplement during the Screening Phase, or is not willing or able to abide by the restrictions regarding use of prohibited medications or dietary supplements;
14. Reports using prokinetics, metformin, regular or frequent antibiotics, systemic glucocorticosteroids, regular non-steroidal anti-inflammatory drugs, sucralfate, ketoconazole, anticholinergics, or misoprostol. The regular intake of acetylsalicylic acid at doses up to 162 mg/day is permitted.
15. Has used an antimicrobial mouth rinse within 1 month of enrollment (e.g. Listerene, etc.);
16. Having ever taken ISOThrive previously
17. History of recurrent infectious condition that requires intermittent antibiotic use
18. If female, is pregnant, lactating, or intending to become pregnant before, during or within 4 weeks after participating in this study or intending to donate ova during such time period
19. Primary sleep disorder including sleep apnea, restless leg syndrome, or insomnia
20. Colon prep or high colonic within 30 days prior to study entry
21. Use of any investigational product within 90 days prior to study entry
22. Participation in another investigation (clinical trial) during the course of this study
23. Participation in a rigorous weight loss program or have any planned changes in diet or lifestyle, such as getting married, change in residence, change in job, or other highly stressful event at any time during the study
24. Diagnosis of inflammatory bowel disease or chronic diarrhea, although a diagnosis of IBS-C or CIC with intermittent short-term diarrhea is acceptable
25. Employment (or relative of an employee) or involvement in any way with ISOThrive Inc.
26. An investigator, key study personnel or first degree relative of anyone involved with the study
27. Other conditions or situations that, in the investigator's opinion, may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2021-04-02 (Actual); Study Completion 2021-04-02 (Actual)

PRIMARY OUTCOMES:
Tolerability of ISOThrive using Patient Assessment of Constipation Quality of Life Questionnaire (PAC-QOL) | 5 weeks
  PAC-QOL a validated questionnaire which measures subject experience over the prior 2 weeks, includes a total of 28 items in 4 subscales: worries and concerns (11 items), physical discomfort (4 items), psychosocial discomfort (8 items), and satisfaction (5 items). Higher scores of PAC-QOL indicate more negative effects of constipation on the quality of life.
  This study will assess whether subjects with constipation tolerate ISOThrive by measuring the differences in baseline and post-intervention score using PAC-QOL. The score taken at the end of Week 1 of the Screening Phase will be compared to the scores at the end of Week 2 and Week 4 of the Tolerability Phase. Any difference in scores between Week 2 and Week 4 of the Tolerability Phase will also be compared. Tolerability is defined as the difference between the baseline score and the post-intervention score at Week 4 of the Tolerability Phase. It must be equal to or less than the baseline score.
Tolerability of ISOThrive using Patient Assessment of Constipation Symptoms (PAC-SYM) | 5 weeks
  PAC-SYM is a validated 12 item constipation symptom questionnaire assessing symptoms over the prior 2 weeks. Sub-scores and total score vary from 0 to 4. All scores are given equal weight. A lower score indicates less symptom severity.
  This study will assess whether subjects with constipation tolerate ISOThrive by measuring the differences in baseline and post-intervention score using PAC-SYM. The score taken at the end of Week 1 of the Screening Phase will be compared to the scores at the end of Week 2 and Week 4 of the Tolerability Phase. Any difference in scores between Week 2 and Week 4 of the Tolerability Phase will also be compared. Tolerability is defined as the difference between the baseline score and the post-intervention score at Week 4 of the Tolerability Phase. It must be equal to or less than the baseline score.
Tolerability of ISOThrive using the Bristol Stool Scale (BSS) | 5 weeks
  This study will assess whether subjects with constipation tolerate ISOThrive by measuring differences in pre and post-intervention scores using the BSS and bowel movement frequency. Electronic BSS diaries will be recorded daily. The BSS is an indicator of colonic transit time using a seven-point scale. Type 1 and 2 indicate hard stool; type 3, 4 and 5 show looser (ideal) stool; and type 6 and 7 indicate stool that is too loose. Tolerability is primarily defined as an increase in the frequency of bowel movements. Tolerability is secondarily defined as improvement in quality, a larger percentage of scores of 3, 4, and 5. Any difference in scores between weeks 1, 2, 3, and 4 of the Tolerability Phase will also be compared. Tolerability is defined as follows: average week 4 stool quality must be equal to or improved (equal to or more scores of 3, 4 and 5) relative to baseline, and average week 4 bowel movement frequency must be equal to or more than baseline frequency.

SECONDARY OUTCOMES:
Adverse Event Assessment | 5 weeks
  Assess any relevant adverse events

CONTACTS AND LOCATIONS:
Overall Officials: John Selling, MD, Principal Investigator — ISOThrive Inc.
Locations (1):
- ISOThrive Inc., Manassas, Virginia, United States

IPD SHARING:
Plan to Share IPD: No